CLINICAL TRIAL: NCT04378907
Title: Assessing Electronic Cigarette Nicotine Flux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HM20018580; 5U54DA036105-10 (NIH)
Record Dates: First submitted 2020-04-30; First posted 2020-05-07 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Electronic Cigarette Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to determine differences in nicotine delivery, use behavior, (puff topography), and carbon monoxide delivery, subjective effects, and physiological effects, when cigarette smokers use an electronic cigarette with constant device settings and different e-liquid concentrations. Only one arm enrolled.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiemental (Experimental): Only one arm enrolled. ECIG Lab Session, 30 watts . During each session (intervention) participants will first complete a 10-puff product use bout, and then a 90-minute product use bout.
  Interventions: Other: Cigarette Smoker/ECIG users: 0 mg/ml nicotine concentration; Other: Cigarette Smokers/ECIG users: 6 mg/ml nicotine concentration; Other: Cigarette Smokers/ECIG users: 15 mg/ml nicotine concentration; Other: Cigarette Smokers/ECIG users: 30 mg/ml nicotine concentration

INTERVENTIONS:
Other: Cigarette Smoker/ECIG users: 0 mg/ml nicotine concentration — ECIG LAB SESSION: 30 watts, 0 mg/ml nicotine concentration. During each session, participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
Other: Cigarette Smokers/ECIG users: 6 mg/ml nicotine concentration — ECIG Lab Session, 30 watts, 6 mg/ml nicotine concentration. During each session, participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
Other: Cigarette Smokers/ECIG users: 15 mg/ml nicotine concentration — ECIG Lab Session, 30 watts, 15 mg/ml nicotine concentration. During each session, participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
Other: Cigarette Smokers/ECIG users: 30 mg/ml nicotine concentration — ECIG Lab Session, 30 watts, 30 mg/ml nicotine concentration
  During each session, participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.

SUMMARY:
The purpose of this study is to determine differences in nicotine delivery, use behavior, carbon monoxide delivery, subjective effects, and physiological effects, when cigarette smokers use an electronic cigarette with constant device settings and different e-liquid concentrations.

DETAILED DESCRIPTION:
Only one arm enrolled.

ELIGIBILITY:
Inclusion Criteria:

* healthy (determined by self-report)
* between the ages of 18-55
* willing to provide informed consent
* able to attend the lab and abstain from tobacco/nicotine as required and must agree to use designated products according to study protocol

Exclusion Criteria:

• Women if they are breast-feeding or test positive for pregnancy (by urinalysis) at screening.

Some study details about the eligibility criteria are purposely omitted at this time to preserve scientific integrity. Full details will be posted at the conclusion of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Breland, PhD, Study Director — Virginia Commonwealth University
Locations (1):
- Center for the Study of Tobacco Products, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this single-arm study, 33 were enrolled. Participants completed four, approximately 3-hr sessions.
Pre-assignment Details: 33 were enrolled
Groups:
- E-cig/Smokers: There was only one arm enrolled. Participants completed four, approximately 3-hr sessions throughout the study.
  * Session 1: Cigarette Smoker/ECIG users: 0 mg/ml nicotine concentration: 30 watts, 0 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 2: Cigarette Smokers/ECIG users: 6 mg/ml nicotine concentration: 30 watts, 6 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 3: Cigarette Smokers/ECIG users: 15 mg/ml nicotine concentration: Session, 30 watts, 15 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 4: Cigarette Smokers/ECIG users: 30 mg/ml nicotine concentration: 30 watts, 30 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
Period: Overall Study
Arm/Group | E-cig/Smokers
Started | 33
Completed | 32
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Demographic information is reported for the 32 participants who completed the study. Only one arm enrolled.
Groups:
- Cigarette Smokers/ECIG Users: Participants completed four, approximately 3-hr sessions throughout the study.
Arm/Group | Cigarette Smokers/ECIG Users
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] — Only one arm enrolled.
  years | 29.41 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants] — Only one arm enrolled.
  Participants
    Female | 11
    Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Only one arm enrolled.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 31
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Only one arm enrolled.
  Participants
    American Indian or Alaska Native | 0
    Asian | 5
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 5
    White | 17
    More than one race | 2
    Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants] — Only one arm enrolled.
  Participants
    United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Plasma Nicotine Concentration
Description: Blood will be taken during each session (5) to examine changes from baseline to immediately follow a ten-puff bout. There is one arm, but 4 different conditions per outcome. One subject with/ missing plasma samples was removed from analysis.
Time Frame: Before directed bout, after directed bout, prior to ad lib use, after ad lib use, and immediately after own brand use.
Population: One arm enrolled and the subjects received each of the 4 conditions. 1 subject with/ missing plasma samples was removed from analysis.
Measure: Mean (Standard Deviation); unit: mg/ml
Groups:
- Experimental Arm/ 0mg Condition; Experimental Arm/ 6mg Condition; Experimental Arm/ 15 mg Condition; Experimental Arm/ 30mg Condition: There was only one arm enrolled. Participants completed four, approximately 3-hr sessions throughout the study.
  * Session 1: Cigarette Smoker/ECIG users: 0 mg/ml nicotine concentration: 30 watts, 0 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 2: Cigarette Smokers/ECIG users: 6 mg/ml nicotine concentration: 30 watts, 6 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 3: Cigarette Smokers/ECIG users: 15 mg/ml nicotine concentration: Session, 30 watts, 15 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 4: Cigarette Smokers/ECIG users: 30 mg/ml nicotine concentration: 30 watts, 30 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
Arm/Group | Experimental Arm/ 0mg Condition | Experimental Arm/ 6mg Condition | Experimental Arm/ 15 mg Condition | Experimental Arm/ 30mg Condition
Number analyzed (Participants) | 31 | 31 | 31 | 31
mg/ml
  Before directed bout | 2.00 (2.86) | 1.92 (2.59) | 1.64 (2.34) | 1.62 (2.53)
  After directed bout | 1.93 (2.80) | 4.75 (3.44) | 8.80 (7.41) | 12.42 (12.21)
  Before ad lib use | 1.74 (2.36) | 3.29 (2.29) | 5.28 (3.79) | 7.62 (5.75)
  After ad lib use | 1.62 (2.15) | 5.39 (3.32) | 8.61 (7.47) | 11.05 (8.71)
  After own brand use | 10.93 (9.67) | 15.05 (10.04) | 16.55 (10.40) | 17.01 (9.70)

2. Primary Outcome: Cigarette/ECIG Challenge Paradigm
Description: Subjects, following a period of abstinence, they are given a limited time to use either their own brand of cigarette or an e-cigarette. One arm enrolled and the subjects received each of the 4 conditions per outcome.
Time Frame: Completion of ad lib bout to use of own brand cigarette
Population: One arm enrolled and the subjects received each of the four conditions per outcome.
Measure: Mean (Standard Deviation); unit: latency to puff own brand in seconds
Groups:
- Experimental Arm/0 mg Condition; Experimental Arm/6 mg Condition; Experimental Arm/ 15 mg Condition; Experimental Arm/ 30 mg Condition: There was only one arm enrolled. Participants completed four, approximately 3-hr sessions throughout the study.
  * Session 1: Cigarette Smoker/ECIG users: 0 mg/ml nicotine concentration: 30 watts, 0 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 2: Cigarette Smokers/ECIG users: 6 mg/ml nicotine concentration: 30 watts, 6 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 3: Cigarette Smokers/ECIG users: 15 mg/ml nicotine concentration: Session, 30 watts, 15 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 4: Cigarette Smokers/ECIG users: 30 mg/ml nicotine concentration: 30 watts, 30 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
Arm/Group | Experimental Arm/0 mg Condition | Experimental Arm/6 mg Condition | Experimental Arm/ 15 mg Condition | Experimental Arm/ 30 mg Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
latency to puff own brand in seconds | 7.74 (4.59) | 10.18 (12.27) | 10.51 (9.57) | 11.64 (12.10)

3. Secondary Outcome: Puff Volume
Description: Puff volume.
Time Frame: During directed bout, during ad lib bout
Population: 32 subjects started the study procedures and 27 completed this study procedure. One arm enrolled and the subjects received each of the four conditions per outcome.
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Experimental Arm/ 0 mg Condition; Experimental/ 6 mg Condition; Experimental Arm/ 15 mg Condition; Experimental Arm/ 30 mg Condition: There was only one arm enrolled. Participants completed four, approximately 3-hr sessions throughout the study.
  * Session 1: Cigarette Smoker/ECIG users: 0 mg/ml nicotine concentration: 30 watts, 0 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 2: Cigarette Smokers/ECIG users: 6 mg/ml nicotine concentration: 30 watts, 6 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 3: Cigarette Smokers/ECIG users: 15 mg/ml nicotine concentration: Session, 30 watts, 15 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 4: Cigarette Smokers/ECIG users: 30 mg/ml nicotine concentration: 30 watts, 30 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
Arm/Group | Experimental Arm/ 0 mg Condition | Experimental/ 6 mg Condition | Experimental Arm/ 15 mg Condition | Experimental Arm/ 30 mg Condition
Number analyzed (Participants) | 27 | 27 | 27 | 27
ml
  Directed bout | 424.46 (235.73) | 425.48 (248.99) | 363.21 (184.21) | 328.52 (181.95)
  Ad lib bout | 400.87 (220.94) | 372.31 (232.72) | 340.99 (194.09) | 298.76 (185.46)

4. Secondary Outcome: Puff Duration
Description: Puff duration measured in seconds.
Time Frame: During directed bout, during ad lib bout
Population: 32 subjects began the study procedures, only 27 completed the study procedure. The results are reported as a single arm, 4 conditions per outcome.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Experimental Arm/ 6 mg Condition; Experimental Arm/ 15 mg Condition; Experimental Arm/ 30 mg Condition: There was only one arm enrolled. Participants completed four, approximately 3-hr sessions throughout the study.
  * Session 1: Cigarette Smoker/ECIG users: 0 mg/ml nicotine concentration: 30 watts, 0 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 2: Cigarette Smokers/ECIG users: 6 mg/ml nicotine concentration: 30 watts, 6 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 3: Cigarette Smokers/ECIG users: 15 mg/ml nicotine concentration: Session, 30 watts, 15 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  * Session 4: Cigarette Smokers/ECIG users: 30 mg/ml nicotine concentration: 30 watts, 30 mg/ml nicotine concentration. Participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
Arm/Group | Experimental Arm/ 0mg Condition | Experimental Arm/ 6 mg Condition | Experimental Arm/ 15 mg Condition | Experimental Arm/ 30 mg Condition
Number analyzed (Participants) | 27 | 27 | 27 | 27
seconds
  Directed bout | 2.31 (0.46) | 2.32 (0.51) | 2.16 (0.41) | 2.01 (0.52)
  Ad lib bout | 2.26 (0.66) | 2.08 (0.68) | 2.08 (0.57) | 1.91 (0.59)

ADVERSE EVENTS:
Time Frame: Data were collected through the subjects participation during the study intervention visits, an average of 2 months.
Description: Data were collected through the subjects participation during the study intervention visits.
Groups:
- Experimental: ECIG Lab Session, During each session, participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout. ECIG Lab Session, 30 watts: During each session, participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout. There was only one arm enrolled and the all of the subjects received the different concentrations in the same order
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT04378907/Prot_001.pdf
  • Informed Consent Form (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT04378907/ICF_000.pdf